CLINICAL TRIAL: NCT02081170
Title: The Intravitreal Autologous Platelet Concentrate Injection as an Adjunct of Vitrectomy for the Treatment of Refractory Macular Holes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-12-066
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Macular Hole With High Myopia (Spherical Equivalent ≤ -6.0 Diopters) or,; Large Size Macular Hole (Diameter > 600 Microns) or; Recurred or Failed Macular Hole From Previous Surgery; or Chronic Macular Hole (Symptom Duration > 6 Months)
MeSH Terms: conditions — Recurrence

ARMS (1):
- autologous platelet concentrate (Experimental)
  Interventions: Procedure: Autologous platelet concentrate

INTERVENTIONS:
Procedure: Autologous platelet concentrate — 1. pars plana vitrectomy
  2. internal limiting membrane removal
  3. Fluid-air exchange
  4. Intravitreal autologous platelet concentrate injection
  5. Intravitreal gas (14% C3F8) injection
  6. Keep prone position for 7-14 days after surgery

SUMMARY:
The purpose of this study is to determine the effectiveness of intravitreal autologous platelet concentrate (APC) injection during the surgery for refractory macular holes.

ELIGIBILITY:
Inclusion Criteria:

* Macular hole with any of following condition

  * High myopia (spherical equivalent ≤ -6.0 Diopters)
  * Large size macular hole (Diameter > 600 microns)
  * Recurred or failed macular hole from previous surgery
  * Chronic macular hole (symptom duration > 6 months)

Exclusion Criteria:

* Systemic infection
* Hematologic disease
* Severe maculopathy including severe diabetic retinopathy, advanced age-related macular degeneration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
macular hole closure | 6 months

SECONDARY OUTCOMES:
best-corrected visual acuity | 6 months
metamorphopsia score | 6 months
safety outcome | 6 months
  frequency and severity of ocular adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea